CLINICAL TRIAL: NCT05709405
Title: Reading Instruction for Children With Intellectual Disabilites Who Require Augmentative and Alternative Communication: a Multiple Random Baselines Design
Brief Title: Reading Intervention for Children With Intellectual Disabilities Who Require Augmentative and Alternative Communication
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Collaborators: University of South-Eastern Norway (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 988724
Record Dates: First submitted 2023-01-10; First posted 2023-02-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Intellectual Disabilities
Keywords: Intellectual disabilities; AAC; Reading intervention; Sound blending; Letter-sound correspondence; Phoneme segmentation; Shared reading; Sight words; Decoding
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Multiple random baseline design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reading Intervention (Experimental): The reading material is made based on the research of Professor Janice Light and Professor David McNaughton at Penn State University. The reading material "Lesing for alle" (Reading for all) contains all the principles, strategies, and methods that form the basis of Accessible Literacy Learning (ALL). The intervention is conducted by trained teachers, in a place known to the students. The material contains: tasks in sound blending, letter-sound correspondence, phoneme- segmentation, sight words, single-word decoding, and shared reading.
  Due to the multiple single baseline design, each participant will be regarded as being in the control condition, and then will be randonly assigned to four different baselines starting the intervention individually after the 2nd, 3rd, 4th, and 5th month.
  Interventions: Other: Reading intervention

INTERVENTIONS:
Other: Reading intervention — The intervention will use a reading program called "Lesing for alle" (Reading for all) based on the research of Accessible Literacy Learning (ALL) which is an evidence-based approach, designed to teach reading skills to students with various intellectual disabilities, including autism spectrum disorders

SUMMARY:
The goal of this multiple single case study with multiple randomized baseline (with four starting points and 18 measurements across time) is to conduct a reading intervention for 40 children with intellectual disabilities who require augmentative and alternative communication (AAC).

The main questions to answer are:

1. Is there a functional relation between the use of "Lesing for alle" (Reading for all) and increased accuracy of sound blending by students age 6-14 with intellectual disabilities who require AAC?
2. Is there a functional relation between the use of "Lesing for alle" (Lesing for alle) and improved acquisition of letter sound correspondence by students age 6-14 with intellectual disabilities who require AAC?
3. Is there a functional relation between the use of "Lesing for alle" (Reading for all) and improved acquisition of phoneme segmentation by students age 6-14 with intellectual disabilities who require AAC?
4. Is there a functional relation between the use of "Lesing for alle" (Reading for all) and improved acquisition of recognition of sight words by students age 6-14 with intellectual disabilities who require AAC?
5. Is there a functional relation between the use of "Lesing for alle" (Reading for all) and improved acquisition of decoding by students age 6-14 with intellectual disabilities who require AAC?
6. Is there a positive and strong correlation between increasing skills from 1-3 and 4-5? Meaning, is there a transfer from lower level skills (phonological skills) to decoding skills?

The participants (age 6-14) will receive daily instruction in a reading material that follows all the strategies of Accessible Literacy Learning, developed by Janice Light and David McNaughton. It is the teachers who will carry out the teaching in the students fixed and familiar place at school. The reading material consist of tasks in sound blending, letter-sound correspondence, phoneme segmentation, sight words and decoding. The reading material will use explicit instruction, distributed and cumulative practice, and immediate and corrective feedback. The intervention will take place for a total of 18 months.

DETAILED DESCRIPTION:
The acquisition of reading skills is a critical need for all individuals and allow fuller participations in education and employment and gives access to personal expression, social media and enjoyable leisure pursuits. Individuals with intellectual disabilities who require augmentative and alternative communication (AAC) often face challenges in that they are met with too low expectations and low ambitions. There is also a lack of evidence-based reading programs and reading materials adapted for individuals who require AAC.

This study will conduct a reading intervention for children with intellectual disabilities who require augmentative and alternative communication (AAC). Through the reading intervention, students will work with components such as sound blending, letter-sound correspondence, phoneme segmentation, sight words, shared reading and decoding. It will be used components of effective evidence-based literacy intervention such as explicit instruction, distributed and cumulative practice, and immediate and corrective feedback. All the instructional activities have been adapted, oral/spoken responses are not required, and the students can use alternative methods, such as signs, pointing at symbols or pointing with their eyes.

The aim of this study is to conduct a reading intervention for 40 children with intellectual disabilities who require augmentative and alternative communication (AAC) to see if the students can acquire functional reading skills. Even simple reading skills can contribute to major changes in the individual's quality of life and to a greater independence in communication with the environment.

ELIGIBILITY:
Inclusion Criteria:

* Students between 6 and 14
* Students who are diagnosed with intellectual disabilities
* Students who do not have a functional speech, i.e. require augmentative and alternative communication (AAC) to understand and/or make oneself understood.
* Students must use AAC as their primary form of communication
* Students cannot follow ordinary curricula (LK20) but have their own education plan.

Exclusion Criteria:

* Students younger than six years and older than 14 years
* Students who have not been diagnosed within intellectual disabilities
* Students who have a functional speech and do not require AAC
* Students who follow ordinary education

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-18 (Estimated)

PRIMARY OUTCOMES:
Sound-blending trajectory change | Every month, for 18 months
  Testing in sound blending involves testing the student's ability to combine individual sounds into words. The students will see a sheet of paper with four symbols. In the instructions, the target word will be presented by expanding the individual sound in the word.
Letter-sound correspondence trajectory change | Every month, for 18 months
  Tests the student's ability to associate letter-sounds with corresponding letters. The students must discriminate between 4 symbols, and the instruction is, for example: point to "0".
Phoneme segmentation trajectory change | Every month, for 18 months
  The students are measured on their ability to find the first sound in words. In the test, there must be discrimination between 4 symbols, and students must identify the word that begins with, for example, the sound "m".

SECONDARY OUTCOMES:
Sight-words change | Three time points before, during, and after intervention (months 1, 12 and 18)
  Tests the students ability to recognize words they have learned by sight.
Decoding change | Three time points before, during and after intervention (months 1, 12 and 18)
  Tests the students ability to convert the printed code (letters) of traditional ortography into words in order to derive meaning.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Larsen, Phd, Study Director — University of South-Eastern Norway
Locations (2):
- Norway (2):
  - Østfold University College, Halden, BRA Veien
  - University of South-Eastern Norway, Borre, Vestfold

REFERENCES:
- [Derived] Ulriksen LB, Bilet-Mossige M, Moreira HC, Larsen K, Nordahl-Hansen A. Reading intervention for students with intellectual disabilities without functional speech who require augmentative and alternative communication: a multiple single-case design with four randomized baselines. Trials. 2023 Jun 27;24(1):433. doi: 10.1186/s13063-023-07452-4. PMID 37370125